CLINICAL TRIAL: NCT04951934
Title: Prospective, Randomized Controlled, Multi-center Study on the Reactivation of the Reparative Process and Scarring Outcome, in Patients Treated With the EmoLED Medical Device, With Deep Burns in Which the Autologous Skin Graft Has Failed
Brief Title: Prospective Randomized International Study on the Reactivation of Burn Injuries
Acronym: SPRINT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There has been no unanimous approval by the investigators regarding the approval of the study protocol. Therefore, by mutual agreement, sponsor and investigators have taken the decision to withdraw the clinical study.
Sponsor: Emoled (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EmoLED_Burn_001
Record Dates: First submitted 2021-06-30; First posted 2021-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Burns; Skin Graft (Allograft)(Autograft) Failure
Keywords: Burns; Graft; Autograft; EmoLED; blue light; LED; blue LED; wound healing
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Multi-centric prospective, randomized controlled study
Masking Description: Since this is an experiment with a medical device that emits blue light, in this case the masking of the assignment to one of the two groups cannot be carried out.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EmoLED Group (Experimental): The EmoLED Group will undergo treatment with EmoLED twice a week for 5 consecutive weeks. The therapy, in this case, in addition to the standard treatment, will also include a treatment with the EmoLED device.
  Interventions: Device: EmoLED; Procedure: Standard treatment
- Control Group (Active Comparator): The Control Group will follow the standard treatment indicated.
  Interventions: Procedure: Standard treatment

INTERVENTIONS:
Device: EmoLED — This treatment consists of irradiation with the blue light emitted by the device for one minute on the injured area. If the wound has a greater extension than the irradiated area, multiple repeated applications will be performed on adjacent areas, until the entire wound is covered.
  Arms: EmoLED Group
Procedure: Standard treatment — The standard treatment consists of: cleansing and possible debridement of the wound, application of the topical treatment indicated for that phase of the wound, intended as the "standard of care" of the structure, and subsequent bandaging.
  Other Names: SOC

SUMMARY:
This clinical trial will be a multi-centric prospective, randomized controlled study with the commercial objective of evaluating the clinical efficacy of a battery-powered portable device that uses blue LEDs. The clinical study aims to compare the existing standard treatment for burned areas in which the autologous skin graft was not successful, with a protocol that includes the administration of the treatment with EmoLED for 5 consecutive weeks in addition to conventional therapy.

The enrolled patients will have to be examined after 5 weeks of treatment, until complete healing and subsequently their scarring will have to be evaluated at 3 and 6 months after healing.

DETAILED DESCRIPTION:
Burns are the fourth most common type of trauma in the world, after traffic accidents, falls and personal violence. Around 11 million people worldwide used medical treatment for burns in 2004. The risk of burns increases with the lowering of the socioeconomic status. Of these burn victims, about 2% need hospitalization and about 0.5% need to be hospitalized in specialized centers.

In deep burns, the surgical procedure of autologous skin transplant (autograft) is almost always the preferred way to induce a re-epithelization of the injured area. The coverage of a deep burn with the graft is -depending on the case case- immediate, delayed a few days after excision or late, after a first phase of direct scarring. Numerous are the types of surgery as well as the sites of skin removal.

The autologous graft, however, presents a not negligible probability of failure that leads to the total or partial detachment of the grafted skin; when this happens the healing process of the lesion (or a part of it) uncovered occurs by second intention but is not always easy to manage, as this process can be delayed or stopped by many factors. Known factors contributing to this are, for example, diabetes, infections, metabolic deficiencies and the advanced age of the subject, while others are still being studied.

Therefore, proper wound management and dressing after surgery, trauma or disease is an important part of the healing process, not only to prevent the onset of infections or other complications, but also to accelerate wound healing itself with as little scarring as possible.

This clinical study will be a multi-centric prospective, randomized controlled parallel group, superiority study, with the commercial objective of evaluating the clinical efficacy of a battery-powered portable device that uses blue LEDs. The Study aims, within the planned observation weeks, to clinically compare two groups of patients with deep burn injuries whose autologous skin graft has failed in part or totally. The objective is to determine any differences in outcome between the two groups considered and whether the therapy of the treatment group is a valid alternative to the current therapy in terms of reactivation and support of the reparative process, speed of healing and scarring.

Group 1, the "Control" group, will follow the standard treatment provided by the hospital protocol; Group 2, the "Treated" one, will follow the standard treatment provided by the hospital protocol to which is added the treatment with the EmoLED device, scheduled between the cleansing and the dressing.

The measurement of the difference in efficacy of the device between the two arms will be evaluated in terms of reactivation of the healing process, intended as the achievement of a re-epithelialization of at least 30%, speed (time) of healing and scarring (Vancouver scale).

The clinical trial in question aims, therefore, to investigate whether the group of patients undergoing standard therapy with, in addition, the treatment with EmoLED reaches a higher percentage of reactivations of the healing process than the one of the control group, subjected to standard treatment. If confirmed, this result would imply significant gains in terms of speeding up hospital stay for those patients where autologous grafts have not been successful, therefore also in terms of reducing public health expenditure, not to mention that, if the improvement of scarring results were confirmed in the Treated group, it would increase the quality of life of patients with burn scars which often significantly impact on this parameter.

The population subject of this trial is widely representative of the target population, as there are no particular exclusion criteria and the sites involved are structures of excellence in the treatment of burns and failed skin grafting areas.

ELIGIBILITY:
Inclusion Criteria:

* Subjects suffering from deep burns who have been surgically treated with autologous skin graft, whose failure has been total or partial;
* The surface of the non-taken skin graft must be between 0.5% and 5.0% of the body surface;
* Men and women aged ≥ 18 years;
* The patient must be able to understand the purpose of the Clinical Study and provide their Informed Consent in writing.

Exclusion Criteria:

* Patients who are participating in other clinical trials with drug or medical device;
* Patients who are unable to understand the aims and the objectives of the study;
* Patients with burns with TBSA greater than 50%;
* Patients with a history of self-harm who can voluntarily alter the course of healing;
* Patients with psychiatric disorders;
* Women who are pregnant or breastfeeding (the state of pregnancy or breastfeeding will be certified on the basis of the patient's declaration);
* Patients with cancer;
* Patients with pathologies that induce photosensitization of the skin;
* Patients with limited life expectancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Patient with an at least 30% area reduction | 5 weeks
  Percentage of patients in the two groups who, after 5 weeks of treatment, achieve a percentage reduction in the wound area of at least 30%.

SECONDARY OUTCOMES:
Percentage surface change | 5 weeks
  Percentage of surface reduction of the wound in the five weeks of observation, in the two treatment groups.
Healing time | 6 months
  Time to achieve healing (indended as the complete re-epithelialization of the observed area), in the two treatment groups.
Scarring | 6 months
  Evaluation of the scarring outcome, using the Vancouver Scar Scale (VSS), three and six months after the complete healing, in the two treatment groups. In the Vancouver Scar Scale, which assesses 4 variables (vascularity, height/thickness, pliability, and pigmentation), "0" is the minimum value and the better outcome, and "13" is the maximum value and worse outcome.
Adverse events | 6 months
  Safety of treatment (number of related adverse events in the two groups).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Gasperini, MD, Study Director — Medical Advisor
Locations (6):
- Medical University of Graz - Department of Surgery - Division of Plastic, Reconstructive and Aesthetic Surgery, Graz, Austria
- Italy (5):
  - AO for emergency "Cannizzaro" - Big Burns Center, Catania
  - Plastic Surgery - Centro Ustioni ASL3 Liguria - Hospital Villa Scassi, Genova
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - AO Cardarelli - UOC Big Burns Center - Reconstructive Plastic Surgery, Napoli
  - AOU Pisana - Sede di Cisanello - UO Burns Center, Pisa